CLINICAL TRIAL: NCT07112209
Title: Evaluation of the Efficacy and Safety of Rezvilutamide Combined With Docetaxel in the Treatment of Abiraterone-resistant Prostate Cancer.
Brief Title: Clinical Study of Rezvilutamide Combined With Docetaxel Chemotherapy in the Treatment of Abiraterone-Resistant Prostate Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-KY-203-02
Record Dates: First submitted 2025-07-15; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-06

CONDITIONS: Pathological and Imaging Examinations Confirmed Metastatic Prostate Cancer
Keywords: abiraterone; PCa; Rezvilutamide; drug resistant; docetaxel
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rivelutamide combined with docetaxel and castration therapy (Experimental): Drug:Rivarestatine Description: 240mg, po, qd Drug:Docetaxel Description:75mg/m2，ivgtt q3w Drug:Prednisone Description:5mg,po,bid
  Interventions: Combination Product: Rezvilutamide combined with docetaxel

INTERVENTIONS:
Combination Product: Rezvilutamide combined with docetaxel — Intervention Description:
  Drug:Rivarestatine Description: 240mg, po, qd Drug:Docetaxel Description:75mg/m2，ivgtt q3w Drug:Prednisone Description:5mg,po,bid

SUMMARY:
Emphasize the main 4 points.

1. Trial Name: Evaluate the efficacy and safety of Rezvilutamide combined with docetaxel in the treatment of abiraterone-resistant prostate cancer.
2. Inclusion criteria:

   ① Adult males over 18 years old, excluding healthy volunteers.
   * Pathological and imaging confirmed as metastatic prostate cancer, who have been receiving abiraterone and castration therapy but have experienced serological or imaging progression; ③ Agree to receive Rezvilutamide combined with docetaxel chemotherapy;

     * ECOG score of 0-1, with a physical condition capable of tolerating chemotherapy; ⑤ Voluntarily sign the informed consent for the clinical trial.

   Exclusion criteria:
   * Having other tumor diseases that require treatment;

     * Having a history of epilepsy or any condition that may cause an epileptic seizure; ③ Having severely impaired liver or kidney function, severe cardiovascular or cerebrovascular diseases, or systemic immune system disorders; ④ Having poor physical condition and being unable to tolerate chemotherapy.
3. ain clinical studies: Rezvilutamide: 240mg (3 tablets) each time, once daily, orally; Androgen deprivation therapy: treated with gonadotropin-releasing hormone analogues or having undergone bilateral orchiectomy; Docetaxel chemotherapy: 75mg/m2 of body surface area by intravenous infusion, once every 3 weeks; simultaneously, oral prednisone was taken twice daily, 5mg each time.
4. The follow-up period is 2 years. Follow-up will be conducted according to the follow-up plan at 1, 3, 6, 9, 12, 16, 18, 21, 24 months after treatment. Patients need to undergo regular examinations (family members and the research supervisor will remind them): 1. General physical examination (height, weight, body temperature, blood pressure, heart rate, pulse, etc.) and important physical sign examination (such as urinary system and other special clinical examinations, etc.).

2. Laboratory tests:

1. Blood routine and urine routine tests;
2. Biochemical tests and liver function tests; 3. Adverse events (AE) and serious adverse events (SAE)

DETAILED DESCRIPTION:
Emphasize the main 4 points.

1. Trial Name: Evaluate the efficacy and safety of Rezvilutamide combined with docetaxel in the treatment of abiraterone-resistant prostate cancer.
2. Inclusion criteria:

   ① Adult males over 18 years old, excluding healthy volunteers.
   * Pathological and imaging confirmed as metastatic prostate cancer, who have been receiving abiraterone and castration therapy but have experienced serological or imaging progression; ③ Agree to receive Rezvilutamide combined with docetaxel chemotherapy;

     * ECOG score of 0-1, with a physical condition capable of tolerating chemotherapy; ⑤ Voluntarily sign the informed consent for the clinical trial.

   Exclusion criteria:
   * Having other tumor diseases that require treatment;

     * Having a history of epilepsy or any condition that may cause an epileptic seizure; ③ Having severely impaired liver or kidney function, severe cardiovascular or cerebrovascular diseases, or systemic immune system disorders; ④ Having poor physical condition and being unable to tolerate chemotherapy.
3. ain clinical studies: Rezvilutamide: 240mg (3 tablets) each time, once daily, orally; Androgen deprivation therapy: treated with gonadotropin-releasing hormone analogues or having undergone bilateral orchiectomy; Docetaxel chemotherapy: 75mg/m2 of body surface area by intravenous infusion, once every 3 weeks; simultaneously, oral prednisone was taken twice daily, 5mg each time.
4. The follow-up period is 2 years. Follow-up will be conducted according to the follow-up plan at 1, 3, 6, 9, 12, 16, 18, 21, 24 months after treatment. Patients need to undergo regular examinations (family members and the research supervisor will remind them): 1. General physical examination (height, weight, body temperature, blood pressure, heart rate, pulse, etc.) and important physical sign examination (such as urinary system and other special clinical examinations, etc.).

2. Laboratory tests:

1. Blood routine and urine routine tests;
2. Biochemical tests and liver function tests; 3. Adverse events (AE) and serious adverse events (SAE)

ELIGIBILITY:
Inclusion Criteria:

* Adult males over 18 years old, excluding healthy volunteers. ② Pathological and imaging confirmed as metastatic prostate cancer, who have been receiving abiraterone and castration therapy but have experienced serological or imaging progression; ③ Agree to receive Rezvilutamide combined with docetaxel chemotherapy;

  * ECOG score of 0-1, with a physical condition capable of tolerating chemotherapy; ⑤ Voluntarily sign the informed consent for the clinical trial.

Exclusion Criteria:

* Having other tumor diseases that require treatment;

  * Having a history of epilepsy or any condition that may cause an epileptic seizure; ③ Having severely impaired liver or kidney function, severe cardiovascular or cerebrovascular diseases, or systemic immune system disorders; ④ Having poor physical condition and being unable to tolerate chemotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult males over the age of 18
Enrollment: 20 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2027-06-10 (Estimated); Study Completion 2027-11-06 (Estimated)

PRIMARY OUTCOMES:
PSA response rate | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical University, Guangzhou, Guangdong, China